CLINICAL TRIAL: NCT05293301
Title: Utilization of a Periodontal Endoscope in Nonsurgical Periodontal Therapy: A Randomized, Split-Mouth Clinical Trial
Brief Title: Utilization of a Periodontal Endoscope in Nonsurgical Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB#9587
Record Dates: First submitted 2022-02-10; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Periodontitis, Adult
Keywords: periodontitis; scaling, subgingival; Non-surgical periodontal therapy
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis

STUDY DESIGN:
Intervention Model Description: prospective, randomized, split-mouth, single blinded
Who Masked: Outcomes Assessor
Masking Description: Follow up re-evaluation visits were performed by the same resident ~1month, 3 months, 6 months, and 1 year, who was blinded to lknowing which side of the mouth recieved what type of deep cleaning treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Periodontal Endosccope (Experimental): One randomly assigned side of the mouth received deep cleaning treatment with the operator using a periodontal endoscope or Perioscopy® for magnification
  Interventions: Device: Use of Periodontal Endoscope (Perioscopy®) to enhance visualization while performing teeth deep cleaning
- Traditional Loupes (Active Comparator): One randomly assigned side of the mouth received deep cleaning treatment with the operator using traditional loupe magnification
  Interventions: Device: Use of traditional loupes to enhance magnification to enhance visualization while performing teeth deep cleaning

INTERVENTIONS:
Device: Use of Periodontal Endoscope (Perioscopy®) to enhance visualization while performing teeth deep cleaning — Deep cleaning or scaling and root planing (SRP) using a Periodontal Endoscope or Perioscopy® for enhanced visualization, on teeth in one half of the mouth
  Arms: Periodontal Endosccope
Device: Use of traditional loupes to enhance magnification to enhance visualization while performing teeth deep cleaning — Deep cleaning or scaling and root planing (SRP) using tradional loupes for enhanced visualization on teeth, in the other half of the mouth
  Arms: Traditional Loupes

SUMMARY:
The purpose of this study was to compare the clinical outcomes of teeth deep cleaning or scaling and root planing (SRP) using a periodontal endoscope (Perioscopy®) versus traditional SRP using magnifying loupes for up to twelve months, utilizing a split mouth design.

DETAILED DESCRIPTION:
Twenty-five (25) patients were recruited for the study that exhibited mild to moderate periodontitis. SRP or deep cleaning was rendered by the same experienced hygienist, following random assignment of the left or right half of the mouth to either recieve deep cleaning by using a periodontal endoscope (Perioscopy®) or traditional deep cleaning using magnifying loupes. All the periodontal evaluations were done by the same periodontal resident at baseline, one month, three months, six months, and twelve months after deep cleaning.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* in good general health
* given a diagnosis of mild-moderate generalized chronic periodontitis per the 1999 world workshop classification of periodontal diseases and conditions
* required whole mouth SRP
* teeth had a maximum of 6mm probing pocket depth at any site
* at least one molar present in each arch, excluding third molars.

Exclusion Criteria:

* any requirement for antibiotic premedication prior to dental treatment
* uncontrolled hypertension
* uncontrolled diabetes
* subject unwilling to sign the informed consent
* subject needed any antibiotic intervention for unrelated conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Percentage of periodontal sites that improved following use of loupes vs perioscopy from baseline - clinical attachment level in mm | 3 months
  Clinical attachment level (in mm) will be measured at six sites per tooth on all teeth per patient.
Percentage of periodontal sites that improved following use of loupes vs perioscopy from baseline - probing pocket depth in mm. | 3 months
  Probing pocket depth (in mm) will be measured at six sites per tooth on all teeth per patient.
Percentage of periodontal sites that improved following use of loupes vs perioscopy from baseline - presence or absence of bleeding on probing. | 3 months
  The presence or absence of bleeding on probing will be meaured at six sites per tooth on all teeth per patient.
Percentage of periodontal sites that improved following use of loupes vs perioscopy from baseline - clinical attachment level in mm. | 6 months
  Clinical attachment level (in mm) will be measured at six sites per tooth on all teeth per patient.
Percentage of periodontal sites that improved following use of loupes vs perioscopy from baseline - probing pocket depth in mm. | 6 months
  Probing pocket depth (in mm) will be measured at six sites per tooth on all teeth per patient.
Percentage of periodontal sites that improved following use of loupes vs perioscopy from baseline - presence or absence of bleeding on probing. | 6 months
  The presence or absence of bleeding on probing will be meaured at six sites per tooth on all teeth per patient.
Percentage of periodontal sites that improved following use of loupes vs perioscopy from baseline - clinical attachment level in mm. | 12 months
  Clinical attachment level (in mm) will be measured at six sites per tooth on all teeth per patient.
Percentage of periodontal sites that improved following use of loupes vs perioscopy from baseline - probing pocket depth in mm. | 12 months
  Probing pocket depth (in mm) will be measured at six sites per tooth on all teeth per patient.
Percentage of periodontal sites that improved following use of loupes vs perioscopy from baseline - presence or absence of bleeding on probing. | 12 months
  The presence or absence of bleeding on probing will be meaured at six sites per tooth on all teeth per patient.

SECONDARY OUTCOMES:
Comparison of clinical measures of periodontal status of teeth (probing pocket depth) of subgroups of teeth following treatment with loupes vs perioscopy. | 3 months
  Probing pocket depth (in mm) around teeth, will be compared between similar sites on different teeth, including; single-rooted vs multi-rooted teeth, maxillary vs mandibular teeth.
Comparison of clinical measures of periodontal status of teeth (clinical attachment level) of subgroups of teeth following treatment with loupes vs perioscopy. | 3 months
  Clinical attachment level (in mm) around teeth, will be compared between similar sites on different teeth, including; single-rooted vs multi-rooted teeth, maxillary vs mandibular teeth.
Comparison of clinical measures of periodontal status of teeth (bleeding on probing) of subgroups of teeth following treatment with loupes vs perioscopy. | 3 months
  Presence or absence of bleeding on probing around teeth, will be compared between similar sites on different teeth, including; single-rooted vs multi-rooted teeth, maxillary vs mandibular teeth.
Comparison of clinical measures of periodontal status of teeth (probing pocket depth) of subgroups of teeth following treatment with loupes vs perioscopy. | 6 months
  Probing pocket depth (in mm) around teeth, will be compared between similar sites on different teeth, including; single-rooted vs multi-rooted teeth, maxillary vs mandibular teeth.
Comparison of clinical measures of periodontal status of teeth (clinical attachment level) of subgroups of teeth following treatment with loupes vs perioscopy. | 6 months
  Clinical attachment level (in mm) around teeth, will be compared between similar sites on different teeth, including; single-rooted vs multi-rooted teeth, maxillary vs mandibular teeth.
Comparison of clinical measures of periodontal status of teeth (bleeding on probing) of subgroups of teeth following treatment with loupes vs perioscopy. | 6 months
  Presence or absence of bleeding on probing around teeth, will be compared between similar sites on different teeth, including; single-rooted vs multi-rooted teeth, maxillary vs mandibular teeth.
Comparison of clinical measures of periodontal status of teeth (probing pocket depth) of subgroups of teeth following treatment with loupes vs perioscopy. | 12 months
  Probing pocket depth around teeth, will be compared between similar sites on different teeth, including; single-rooted vs multi-rooted teeth, maxillary vs mandibular teeth.
Comparison of clinical measures of periodontal status of teeth (clinical attachment level) of subgroups of teeth following treatment with loupes vs perioscopy. | 12 months
  Clinical attachment level (in mm) around teeth, will be compared between similar sites on different teeth, including; single-rooted vs multi-rooted teeth, maxillary vs mandibular teeth.
Comparison of clinical measures of periodontal status of teeth (bleeding on probing) of subgroups of teeth following treatment with loupes vs perioscopy. | 12 months
  Presence or absence of bleeding on probing around teeth, will be compared between similar sites on different teeth, including; single-rooted vs multi-rooted teeth, maxillary vs mandibular teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mayer, RDH,MS, Principal Investigator — LSUHSC SCHOOL OF DENTISTRY (DEPT. OF PERIODONTICS)
Locations (1):
- LSU Health New Orleans School of Dentistry (Dept of Periodontics), New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No